CLINICAL TRIAL: NCT02776722
Title: The Effect of 'Catalytic' Doses of Fructose and Its Epimers on Acute Postprandial Carbohydrate Metabolism and Longterm Glycemic Control: A Series of Systematic Reviews and Meta-analyses of Controlled Feeding Trials
Brief Title: Meta-analyses of the Effect of 'Catalytic' Doses of Fructose and Its Epimers on Carbohydrate Metabolism
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Canadian Diabetes Association (Other); The Physicians' Services Incorporated Foundation (Other); Banting & Best Diabetes Centre (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, John Sievenpiper, Associate Professor, University of Toronto
Other Study IDs: UT-Fructose epimers
Record Dates: First submitted 2016-05-14; First posted 2016-05-18 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Overweight; Obesity; Dysglycemia; Prediabetes; Metabolic Syndrome; Type 2 Diabetes
Keywords: Systematic Review and Meta-analysis; randomized controlled trial; Evidence-Based Medicine; carbohydrate metabolism; postprandial; glycemic response; glycemic control; insulin sensitivity; beta-cell function; sugars; fructose; allulose; tagatose; sorbose
MeSH Terms: conditions — Overweight; Obesity; Prediabetic State; Metabolic Syndrome; Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Fructose; psicose; tagatose; Sorbose

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: fructose, allulose, tagatose, or sorbose — Single-bolus feeding of fructose, allulose, tagatose, or sorbose given together with a reference carbohydrate(s) compared with the same reference carbohydrate(s) alone for acute feeding trials or chronic feeding of fructose, allulose, tagatose, or sorbose provided in substitution for other reference carbohydrates or added to a control diet compared with the reference carbohydrate(s) alone or the control diet alone for chronic feeding trials.

SUMMARY:
Despite advances in the prevention and treatment of type 2 diabetes, its prevalence continues to rise worldwide. There is a need for new modalities to improve metabolic control in individuals with type 2 diabetes and those who are overweight or obese and at risk for type 2 diabetes. Contrary to the concerns raised about the adverse role of fructose in metabolic health, various lines of evidence suggest that fructose and its epimers may improve the metabolic handling of glucose through inducing glycogen synthesis. Recent small trials in humans suggest that catalytic doses (=<10g/meal) of fructose and its epimers (allulose, tagatose, and sorbose) may reduce postprandial glycemic responses to carbohydrate loads (i.e., oral glucose tolerance test or a starch load) in people with and without type 2 diabetes. There is also limited evidence that these acute effects may manifest as longer term improvements in glycemic control. There is an urgent need to synthesize the evidence of the effects of fructose and its epimers on postprandial carbohydrate metabolism.

DETAILED DESCRIPTION:
Background: Despite advances in the prevention and treatment of type 2 diabetes, its prevalence continues to rise worldwide. There is a need for new modalities to improve glycemic control in individuals with type 2 diabetes and those who are overweight or obese and at risk for type 2 diabetes. Contrary to the concerns raised about the adverse role of fructose in metabolic health, there may be a role for fructose and its epimers, the rare non caloric sugars allulose (C-3 epimer of fructose), tagatose (C-4 epimer of fructose), and D-sorbose (C-3 and C-4 diastereomer of fructose). All are naturally found in small quantities in dried fruits and maple syrup. Bother allulose and tagatose are generally recognized as safe (GRAS) by the Food and Drug Administration in the US and are marketed as low-calorie sugar substitutes that have anti-hyperglycemic effects. Various lines of evidence suggest that fructose and its epimers may improve the metabolic handling of glucose through inducing glycogen synthesis. Recent small trials in humans suggest that 'catalytic' doses (=<10g/meal) of fructose and its epimers (allulose, tagatose, and sorbose) may reduce postprandial glycemic responses to carbohydrate loads (i.e., oral glucose tolerance test or a starch load) in people with and without type 2 diabetes. These acute effects have been shown to be sustainable over the longer term in several controlled trials of fructose and tagatose.

Need for a review: There is an urgent need to synthesize the evidence of the effects of fructose and its epimers on acute postprandial carbohydrate metabolism and longterm glycemic control. There remains uncertainty in regards to the minimum effective dose (range studied, 2-25g) and the extent to which these benefits translate into meaningful longterm improvements in glycemic control. A systematic review and meta-analysis remains the "Gold Standard" of evidence to support health claims development. It will map the available evidence and, by pooling the totality of that evidence, provide the most precise estimate of the true effect of fructose and its epimers on carbohydrate metabolism and longterm glycemic control.

Objectives: The investigators will conduct two systematic reviews and meta-analyses of the effect of small 'catalytic' doses of fructose and its epimers. The objective of the first systematic review and meta-analysis will be to assess their effect on the postprandial glycemic and insulinemic responses to other carbohydrates in acute feeding trials, while the objective of the second systematic review and meta-analysis will be to update and expand on our previous systematic review and meta-analysis of small catalytic doses of fructose to assess the effect of small catalytic doses of fructose and its epimers on glycemic control in chronic feeding trials.

Design: The planning and conduct of the two proposed systematic reviews and meta-analyses will follow the Cochrane handbook for systematic reviews of interventions. The reporting will follow the Preferred Reporting Items for Systematic reviews and Meta-Analyses (PRISMA) guidelines.

Data sources: MEDLINE, EMBASE and The Cochrane Central Register of Controlled Trials will be searched using appropriate search terms.

Study selection: The first systematic review and meta-analysis will include single-bolus feeding trials assessing the effect of small 'catalytic doses (=<10g/meal) of fructose and its epimers on the acute postprandial glycemic and insulinemic responses to other carbohydrates. The second systematic review and meta-analysis will include controlled feeding trials of >=1-week diet duration investigating the effect of small 'catalytic doses (=<50g/day or =<10% energy/day) of fructose and its epimers on markers of glycemic control. The 50g/day =<10% energy/day dose threshold for chronic feeding allows for the intake of fructose and its epimers as part of 3 main meals (=<10g/meal) and 3 snacks (=<5g/meal) per day and aligns with current guidelines not to exceed 10% energy from free or added sugars.

Data extraction: Two or more investigators will independently extract relevant data and assess risk of bias using the Cochrane Risk of Bias Tool. All disagreements will be resolved by consensus. Mean values and SEs will be extracted for all outcomes. Standard computations and imputations will be used to derive missing data.

Outcomes: Acute glycemic outcomes (incremental area under the curve (iAUC) for blood glucose and insulin, Matsuda insulin sensitivity index, and the early insulin secretion index) will be assessed in the first systematic review and meta-analysis while chronic glycemic outcomes (HbA1c, fasting glucose, and fasting insulin) will be assessed in the second systematic review and meta-analysis.

Data synthesis: Ratios of means will be pooled for the acute glycemic outcomes and mean differences will be pooled for the chronic glycemic outcomes using the Generic Inverse Variance method with random effects models. Random-effects models will be used even in the absence of statistically significant between-study heterogeneity, as they yield more conservative summary effect estimates in the presence of residual heterogeneity. Fixed-effects models will only be used where there is <5 included studies. Paired analyses will be applied for crossover trials. Heterogeneity will be tested (Cochran Q statistic) and quantified (I2 statistic). To explore sources of heterogeneity, the investigators will conduct sensitivity analyses, in which each study is systematically removed. If there are >=10 studies, then the investigators will also explore sources of heterogeneity by a priori subgroup analyses by participant phenotype, dose, comparator, baseline measurements, risk of bias, study design (parallel, crossover), energy balance (positive, neutral, negative), and duration of follow-up. Metaregression will assess the significance of categorical subgroup analyses and model continuous dose response relationships. Where no evidence of a linear relationship is observed, meta-regression spline curve modeling will be undertaken (the MKSPLINE procedure) to assess a dose threshold by characterizing segments of the dose-response curve where separate linear approximations may best describe the data. If there are more than 10 trial comparisons, then Publication publication bias will be assessed by inspection of funnel plot and the Egger and Begg tests. If publication bias is suspected, then an adjustment for funnel plot asymmetry will be attempted by imputing the missing study data using the Duval and Tweedie trim-and-fill method.

Evidence Assessment: The strength of the evidence for each outcome will be assessed using the Grading of Recommendations Assessment, Development and Evaluation (GRADE).

Knowledge translation plan: Results will be disseminated through traditional means such as interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Innovative means such as webcasts with e-mail feedback mechanisms will also be used. Knowledge Users will act as knowledge brokers networking among opinion leaders and different adopter groups to increase awareness at each stage. Four Knowledge Users will also participate directly as members of nutrition guidelines committees. Target adopters will include industry and research communities. Feedback will be incorporated and used to guide analyses and improve key messages at each stage.

Significance: The proposed project will aid in knowledge translation related to the effects of fructose and its epimers on postprandial carbohydrate metabolism. This project aims to inform future design of single-meal feeding trials on fructose and its epimers by establishing the dose range for their effects on postprandial carbohydrate metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Controlled trials in humans
* Acute single-bolus feeding of fructose, allulose, tagatose, or sorbose (>=2-hour profile) or chronic feeding of fructose, allulose, tagatose, or sorbose (>= 2-weeks diet duration)
* Doses of fructose, allulose, tagatose, or sorbose of =<10g/meal for acute feeding trials or =<40g/day for chronic feeding trials
* Adequate comparator (reference carbohydrate or control diet)
* Outcome data reported

Exclusion Criteria:

* Non-human studies
* observational studies
* Lack of adequate comparator or control group
* Doses of fructose, allulose, tagatose, or sorbose providing >10g/meal for acute feeding trials or >40g/day for chronic feeding trials
* Follow-up <2-hours for acute feeding trials or < 2-weeks (diet duration) for chronic feeding trials
* Lack of reported outcome data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All individuals, both children and adults, regardless of health status.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Acute glycemic outcome - glycemic response | Up to 20 years
  Incremental area under the curse (iAUC) blood glucose
Acute glycemic outcome - insulinemic response | Up to 20 years
  Incremental area under the curse (iAUC) blood insulin
Acute glycemic outcome - whole body insulin sensitivity | Up to 20 years
  Matsuda whole body insulin sensitivity index
Acute glycemic outcome - beta cell function | Up to 20 years
  Early Insulin Secretion Index
Chronic glycemic outcome - HbA1c | Up to 20 years
  HbA1c
Chronic glycemic outcome - fasting glucose | Up to 20 years
  Fasting blood glucose
Chronic glycemic outcome - fasting insulin | Up to 20 years
  Fasting blood insulin

CONTACTS AND LOCATIONS:
Overall Officials: John Sievenpiper, MD, PhD, FRCPC, Principal Investigator — University of Toronto
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Wu T, Zhao BR, Bound MJ, Checklin HL, Bellon M, Little TJ, Young RL, Jones KL, Horowitz M, Rayner CK. Effects of different sweet preloads on incretin hormone secretion, gastric emptying, and postprandial glycemia in healthy humans. Am J Clin Nutr. 2012 Jan;95(1):78-83. doi: 10.3945/ajcn.111.021543. Epub 2011 Dec 7. PMID 22158727
- [Background] Hayashi N, Iida T, Yamada T, Okuma K, Takehara I, Yamamoto T, Yamada K, Tokuda M. Study on the postprandial blood glucose suppression effect of D-psicose in borderline diabetes and the safety of long-term ingestion by normal human subjects. Biosci Biotechnol Biochem. 2010;74(3):510-9. doi: 10.1271/bbb.90707. Epub 2010 Mar 7. PMID 20208358
- [Background] Iida T, Kishimoto Y, Yoshikawa Y, Hayashi N, Okuma K, Tohi M, Yagi K, Matsuo T, Izumori K. Acute D-psicose administration decreases the glycemic responses to an oral maltodextrin tolerance test in normal adults. J Nutr Sci Vitaminol (Tokyo). 2008 Dec;54(6):511-4. doi: 10.3177/jnsv.54.511. PMID 19155592
- [Background] Donner TW, Wilber JF, Ostrowski D. D-tagatose, a novel hexose: acute effects on carbohydrate tolerance in subjects with and without type 2 diabetes. Diabetes Obes Metab. 1999 Sep;1(5):285-91. doi: 10.1046/j.1463-1326.1999.00039.x. PMID 11225640
- [Background] Kwak JH, Kim MS, Lee JH, Yang YJ, Lee KH, Kim OY, Lee JH. Beneficial effect of tagatose consumption on postprandial hyperglycemia in Koreans: a double-blind crossover designed study. Food Funct. 2013 Aug;4(8):1223-8. doi: 10.1039/c3fo00006k. PMID 23760573